CLINICAL TRIAL: NCT01834872
Title: Safety and Feasibility of Arrhythmia Ablation Using the Amigo Remote Robotic System as Compared With Manual Ablation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Sanitaria Gregorio Marañón (Other)
Collaborators: Catheter Robotics, Inc. (Industry)
Responsible Party: Principal Investigator, Tomas Datino, Dr., Instituto de Investigación Sanitaria Gregorio Marañón
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Arenal - 001
Record Dates: First submitted 2013-04-04; First posted 2013-04-18 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amigo (Experimental): Ablation completed with Amigo
  Interventions: Device: Amigo
- Manual (Active Comparator): Ablation completed with manual catheter
  Interventions: Device: Manual ablation

INTERVENTIONS:
Device: Amigo
  Arms: Amigo
Device: Manual ablation
  Arms: Manual

SUMMARY:
The aim of this prospective observational study is to evaluate the performance of Amigo RCS in ablation procedures for most common arrhythmias as compared to a conventional manual approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to our electrophysiology laboratory to treat any type of arrhythmia with catheter ablation

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Ablation Success | 1 year
  Global efficacy:
  Recurrence rate Re-do procedures Proportion of patients under anti arrhythmic treatment
Safety Endpoint | 1 Year
  Any complications that could be attributed to the procedure during follow-up.

SECONDARY OUTCOMES:
Acute Ablation Success | During Procedure
  Accessory pathway: Anterograde and retrograde conduction block through the accessory Pathway Atrial fibrillation: % patients with all PV disconnected circumferential ablation with electrical disconnection of all pulmonary veins Common-type atrial flutter: Bidirectional cavotricuspid isthmus block AVNRT/Ventricular tachycardia/other atrial arrhythmias: Arrhythmia termination / absence o induction
Acute Safety Endpoint | During Procedure
  Procedure complications: Any complication during the electrophysiological procedure and 1 week post ablation that could be attributed to the procedure: Vascular complication, pericardial effusion/cardiac tamponade, heart failure, others.
  The number of adverse events will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

REFERENCES:
- [Derived] Datino T, Arenal A, Pelliza M, Hernandez-Hernandez J, Atienza F, Gonzalez-Torrecilla E, Avila P, Bravo L, Fernandez-Aviles F. Comparison of the safety and feasibility of arrhythmia ablation using the Amigo Robotic Remote Catheter System versus manual ablation. Am J Cardiol. 2014 Mar 1;113(5):827-31. doi: 10.1016/j.amjcard.2013.11.030. Epub 2013 Dec 12. PMID 24440330